CLINICAL TRIAL: NCT06327230
Title: The Application of Thoracic Epidural Analgesia in Patients With Acute Pancreatitis: A Prospective, Multicenter, Randomized, Parallel-Controlled Clinical Study
Brief Title: The Application of Thoracic Epidural Analgesia in Patients With Acute Pancreatitis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SRRSH2023-0627
Record Dates: First submitted 2024-03-05; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Acute Pancreatitis
MeSH Terms: conditions — Pancreatitis | interventions — Tea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Non-TEA group" (No Intervention): After enrollment, the subjects are given standard treatment, including continuous monitoring of vital signs, pain control with intravenous non-steroidal anti-inflammatory drugs (such as ibuprofen) and intravenous opioids (such as tramadol), goal-directed intravenous fluid resuscitation, correction of electrolyte and metabolic disturbances, nutritional support, use of antibiotics and sedatives as needed, necessary mechanical ventilation, continuous renal replacement therapy (CRRT) and other organ support therapies as needed.
- TEA group (Experimental): Patient in lateral position, standard disinfection, puncture point selected at T7-T9 level, local anesthesia to pierce skin. Direct/lateral needle approach cautiously, confirm entry into epidural space with disappearance of resistance and negative pressure. Insert epidural catheter 3-5cm towards head, secure firmly. Test dose with 3mL 1% lidocaine injection to confirm epidural anesthesia efficacy and safety. Epidural infusion of 0.15% ropivacaine (250mL) + fentanyl (2.5mg) via patient-controlled pump at 5mL/h with bolus option. Adjust infusion rate 1-3mL/h based on pain needs.
  Interventions: Procedure: Thoracic Epidural Analgesia

INTERVENTIONS:
Procedure: Thoracic Epidural Analgesia — Thoracic epidural analgesia is performed by a standardized anesthesia team. Patients are positioned in the lateral decubitus position, and routine disinfection is performed. The puncture site is selected at the T7-T9 level. When encountering sudden disappearance of resistance and appearance of negative pressure during needle advancement, it is determined that the needle has entered the epidural space. After confirming needle tip placement in the epidural space with a test dose, an epidural catheter is inserted approximately 3-5cm cephalad and securely fixed in place. The test dose consists of 3 mL of 1% lidocaine injection solution, administered to observe the level of anesthesia, confirming the effectiveness and safety of the epidural anesthesia. Subsequently, a maintenance regimen of 0.15% ropivacaine 250mL with 2.5mg of hydroma.
  Arms: TEA group

SUMMARY:
Acute pancreatitis (AP) is one of the most common diseases of the digestive system, with its incidence increasing year by year. 15%-25% of patients will develop severe acute pancreatitis (SAP), characterized by necrosis and infection of the pancreas and surrounding tissues, as the investigators as multiple organ dysfunction syndrome (MODS), with a mortality rate as high as 17%. Currently, there is a lack of effective measures in clinical practice to regulate the early inflammation and immune response in acute pancreatitis. Animal experimental studies have confirmed that TEA, by blocking the abdominal sympathetic nerves, increases arterial blood flow and venous capacity, improves pancreatic perfusion insufficiency caused by AP, and alleviates metabolic acidosis. Simultaneously, TEA can suppress the secretion of catecholamines during the stress state of acute pancreatitis, reducing the release of inflammatory mediators and thereby inhibiting the inflammatory response. Our team's earlier animal experiments have further confirmed that TEA improves intestinal inflammation in mice with pancreatitis. This improvement is marked by a significant reduction in the concentrations of inflammatory cytokines such as IL-1β and TNF-α. Additionally, there is an observed alteration in the intestinal microbiota, characterized by an increase in the proportion of beneficial bacteria. Based on these findings, it is speculated that TEA, by reducing catecholamine release and downregulating sympathetic activity, effectively mitigates inflammation and stress responses in patients with pancreatitis. Furthermore, TEA dilates small arteries in blocked segments, thereby improving blood flow and microcirculation within the affected area. Indirectly, TEA increases vagal nerve activity, which in turn slows down the progression of intestinal ischemia, consequently reducing the impact of the "second hit" caused by the translocation of intestinal bacteria and endotoxins into the bloodstream, which exacerbates acute pancreatitis. Despite these promising results, clinical data on the efficacy of TEA in acute pancreatitis remains insufficient. Moreover, the precise mechanisms by which TEA influences the progression and severity of acute pancreatitis are yet to be fully elucidated. In order to further validate the clinical therapeutic effects of TEA and gain a deeper understanding of its mechanisms, the investigators have conducted this clinical study.

DETAILED DESCRIPTION:
Acute pancreatitis (AP) is one of the most common diseases of the digestive system, with its incidence increasing year by year. 15%-25% of patients will develop severe acute pancreatitis (SAP), characterized by necrosis and infection of the pancreas and surrounding tissues, as the investigators as multiple organ dysfunction syndrome (MODS), with a mortality rate as high as 17%. This poses a serious threat to public health and also imposes a heavy burden on medical resources. Further improving the treatment level of acute pancreatitis (especially severe cases) is an urgent problem that needs to be addressed.

Acute pancreatitis is a systemic disease. In the early stages of onset, along with local inflammation in the pancreas, there is a release of a large number of inflammatory mediators, leading to systemic inflammatory response syndrome (SIRS). This can subsequently affect multiple systems including respiratory, circulatory, urinary, digestive, and nervous systems, with severe cases leading to multiple organ dysfunction syndrome (MODS). The necrosis and infection of the pancreas and surrounding tissues can lead to a series of local and systemic complications. It has been confirmed that necrosis, infection, and organ dysfunction are the main reasons for the poor prognosis of pancreatitis. During the acute phase of pancreatitis, systemic inflammatory cells become excessively activated and release large amounts of cytokines, triggering a cascade reaction of inflammatory mediators, leading to systemic inflammatory response syndrome (SIRS) and subsequently inducing multiple organ dysfunction syndrome (MODS). The release of inflammatory factors also leads to damage to the intestinal mucosal barrier, allowing harmful substances or bacteria to pass through the damaged intestinal mucosal barrier into the bloodstream or invade other organs outside the intestines, further exacerbating the development of acute pancreatitis. Following the initial phase of acute inflammation and subsequent translocation of intestinal bacteria and endotoxins into the bloodstream, creating a "second hit," the mortality rate of pancreatitis can reach as high as 10-24%.

Currently, there is a lack of effective measures in clinical practice to regulate the early inflammation and immune response in acute pancreatitis. In recent years, studies have shown that the nervous, endocrine, and immune systems can interact with each other, exerting mutual constraints and playing important roles in the inflammatory stress response6. Thoracic Epidural Anesthesia (TEA) is a commonly used method of nerve blockade in anesthesia. It involves injecting local anesthetic drugs into the epidural space to block the nerve roots, resulting in paralysis of the innervated area. TEA is widely used for postoperative pain management in thoracic and abdominal surgeries. In patients with acute pancreatitis (AP), TEA can block the transmission pathway of visceral sensory pancreatic pain fibers to the brain, thereby reducing the patient's pain and stress response caused by pain, and alleviating the patient's suffering. Low concentrations of local anesthetics can effectively block the sympathetic nerves corresponding to the segment, by reducing sympathetic nerve tension, dilating small arteries in the corresponding segment, and improving blood flow and microcirculation in the blocked area. Animal experimental studies have confirmed that TEA, by blocking the abdominal sympathetic nerves, increases arterial blood flow and venous capacity, improves pancreatic perfusion insufficiency caused by AP, and alleviates metabolic acidosis. Simultaneously, TEA can suppress the secretion of catecholamines during the stress state of acute pancreatitis, reducing the release of inflammatory mediators and thereby inhibiting the inflammatory response. Furthermore, the excessive release of early inflammatory factors in acute pancreatitis (AP) and ischemia-reperfusion injury, among other factors, lead to the release of intestinal bacterial endotoxins into the bloodstream. This triggers a burst release of pro-inflammatory cytokines such as IL-1β and IL-18, which further exacerbates the damage to the intestinal mucosal barrier. Consequently, this imbalance in the microecological environment causes intestinal mucosal edema, erosion, and initiates a vicious cycle of systemic inflammatory response, leading to multi-organ damage and dysfunction. This cycle is a significant contributor to the high mortality and disability rates associated with severe acute pancreatitis. TEA selectively blocks the efferent sympathetic nerve fibers in the thoracic and abdominal segments, indirectly increasing vagal nerve activity. This promotes gastrointestinal motility, improves intestinal blood circulation, slows down the progression of acute intestinal ischemia, and prevents the translocation of intestinal bacteria and endotoxins across the intestinal mucosa. Our team's earlier animal experiments have further confirmed that TEA improves intestinal inflammation in mice with pancreatitis. This improvement is marked by a significant reduction in the concentrations of inflammatory cytokines such as IL-1β and TNF-α. Additionally, there is an observed alteration in the intestinal microbiota, characterized by an increase in the proportion of beneficial bacteria. Based on these findings, it is speculated that TEA, by reducing catecholamine release and downregulating sympathetic activity, effectively mitigates inflammation and stress responses in patients with pancreatitis. Furthermore, TEA dilates small arteries in blocked segments, thereby improving blood flow and microcirculation within the affected area. Indirectly, TEA increases vagal nerve activity, which in turn slows down the progression of intestinal ischemia, consequently reducing the impact of the "second hit" caused by the translocation of intestinal bacteria and endotoxins into the bloodstream, which exacerbates acute pancreatitis. Despite these promising results, clinical data on the efficacy of TEA in acute pancreatitis remains insufficient. Moreover, the precise mechanisms by which TEA influences the progression and severity of acute pancreatitis are yet to be fully elucidated.

In clinical practice, epidural blockade often employs low-concentration local anesthetics combined with opioid medications. Hydromorphone, a semi-synthetic potent opioid, when administered perispinally, not only enhances analgesic effects but also exhibits superior vasodilatory properties compared to other opioids such as epidural morphine and fentanyl. This carries particular clinical significance in improving pancreatic microcirculation in patients with acute pancreatitis (AP).

In this study, the investigators propose employing ropivacaine in combination with hydromorphone for TEA. Our aim is to analyze the inflammatory response and clinical efficacy in patients with acute pancreatitis following the early application of TEA, and to elucidate its protective mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years old (inclusive).
* Admission within 7 days of onset of acute pancreatitis diagnosis.
* Admission to the ICU with single or multiple organ failure (lasting more than 48 hours).
* Voluntary participation in this study and signing of the informed consent form. If the subject is unable to read and sign the informed consent form due to lack of capacity, their legal guardian must participate in the informed consent process and sign the form on their behalf. If the subject is unable to read the informed consent form (e.g., illiterate subjects), a witness must witness the informed consent process and sign the form.

Exclusion Criteria:

* 1.Lactating or pregnant women, or those planning pregnancy within 6 months.
* Chronic pancreatitis or pancreatitis related to pancreatic tumors.
* Previously underwent surgical debridement and drainage.
* Previous cardiopulmonary resuscitation with no neurological recovery.
* History of severe primary cardiovascular, respiratory, renal, hepatic, hematologic, malignant tumor, or immune disease conditions: heart failure patients with New York Heart Association (NYHA) functional class greater than II; active myocardial ischemia undergoing cardiovascular intervention within 60 days.
* Allergy to local anesthetics.
* Anatomical variation preventing "thoracic epidural blockade."
* Coagulation disorders or undergoing anticoagulant therapy.
* Participation in other interventional clinical studies in the past 3 months.
* Other situations deemed unsuitable for inclusion by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
The change in systemic inflammatory response syndrome (SIRS) and organ dysfunction after inclusion. | Day0,1,3,5,7
  SIRS score, APACHE II score, Marshall Organ Dysfunction Score.
The change in intra-abdominal pressure (measured via bladder pressure) after treatment. | day0，"3-6 hours post-treatment"，day1,3,5,7
  obtained from measured data
The change in resting pain and movement pain after inclusion. | day0，"3-6 hours post-treatment"，day1,3,5,7
  When patients are in a state of endotracheal intubation, use the Critical Care Pain Observation Tool (CPOT) for assessment.

SECONDARY OUTCOMES:
Peripheral blood inflammation and immune markers. | From the date of randomization (day 0) and at days 1, 3, 5, and 7.
  Complete Blood Count (CBC)、C-reactive Protein (CRP)、PCT、Epinephrine Levels、T Cell Subpopulation Analysis、IL-6 、IL-10 、TNF-α 、IL-1β etc
intestinal microbiota | From the date of randomization (day 0) and at days 1, 3, 5, and 7.
total ICU treatment time | From the date of randomization until the first documented record of the patient being transferred out of the ICU，assessed up to 6 months
adverse event occurrence rate | From the date of randomization until the first documented occurrence of an adverse event，assessed up to 2 months

CONTACTS AND LOCATIONS:
Overall Officials: hong yu, Principal Investigator — sir run run shaw hospital，hangzhou
Locations (1):
- Sir Run Run Shaw Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No